CLINICAL TRIAL: NCT02573155
Title: A 2-part, Randomised, Placebo-controlled, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of AZD8871 Delivered by Inhalation in Asthmatic and Chronic Obstructive Pulmonary Disease (COPD) Subjects
Brief Title: Two-part Safety, Tolerability, Pharmacodynamic and -Kinetic Study of Inhaled AZD8871 in Asthmatic and COPD Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D6640C00001; 2015-002906-36 (EudraCT Number)
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-04

CONDITIONS: Asthma (Part 1); COPD (Part 2)
Keywords: Pharmacokinetics; Pharmacodynamics; AZD8871; Safety; Tolerability; mild persistent asthma; moderate to severe COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — AZD-8871; indacaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (18):
- Sequence 1, Part 1 (Experimental): Period 1: Dose 1 Period 2: Dose 3 Period 3: Dose 5
  Interventions: Drug: Dose 1, AZD8871 50 μg (Part 1); Drug: Dose 3, AZD8871 300 μg (Part 1); Drug: Dose 5, AZD8871 1200 µg (Part 1)
- Sequence 2, Part 1 (Experimental): Period 1: Placebo Period 2: Dose 3 Period 3: Dose 5
  Interventions: Drug: Dose 3, AZD8871 300 μg (Part 1); Drug: Dose 5, AZD8871 1200 µg (Part 1); Drug: Placebo, AZD8871 placebo (Part 1)
- Sequence 3, Part 1 (Experimental): Period 1: Dose 1 Period 2: Placebo Period 3: Dose 5
  Interventions: Drug: Dose 1, AZD8871 50 μg (Part 1); Drug: Dose 5, AZD8871 1200 µg (Part 1); Drug: Placebo, AZD8871 placebo (Part 1)
- Sequence 4, Part 1 (Experimental): Period 1: Dose 1 Period 2: Dose 3 Period 3: Placebo
  Interventions: Drug: Dose 1, AZD8871 50 μg (Part 1); Drug: Dose 3, AZD8871 300 μg (Part 1); Drug: Placebo, AZD8871 placebo (Part 1)
- Sequence 5, Part 1 (Experimental): Period 1: Dose 2 Period 2: Dose 4 Period 3: Dose 6
  Interventions: Drug: Dose 2, AZD8871 100 μg (Part 1); Drug: Dose 4, AZD8871 600 µg (Part 1); Drug: Dose 6, AZD8871 1800 μg (Part 1)
- Sequence 6, Part 1 (Experimental): Period 1: Placebo Period 2: Dose 4 Period 3: Dose 6
  Interventions: Drug: Dose 4, AZD8871 600 µg (Part 1); Drug: Dose 6, AZD8871 1800 μg (Part 1); Drug: Placebo, AZD8871 placebo (Part 1)
- Sequence 7, Part 1 (Experimental): Period 1: Dose 2 Period 2: Placebo Period 3: Dose 6
  Interventions: Drug: Dose 2, AZD8871 100 μg (Part 1); Drug: Dose 6, AZD8871 1800 μg (Part 1); Drug: Placebo, AZD8871 placebo (Part 1)
- Sequence 8, Part 1 (Experimental): Period 1: Dose 2 Period 2: Dose 4 Period 3: Placebo
  Interventions: Drug: Dose 2, AZD8871 100 μg (Part 1); Drug: Dose 4, AZD8871 600 µg (Part 1); Drug: Placebo, AZD8871 placebo (Part 1)
- Sequence 1, Part 2 (Experimental): Period 1: Treatment A Period 2: Treatment B Period 3: Treatment E Period 4: Treatment C Period 5: Treatment D
  Interventions: Drug: Treatment A, AZD8871 dose A (Part 2); Drug: Treatment B, AZD8871 dose B (Part 2); Drug: Treatment C, Indacaterol 150 μg (Part 2); Drug: Treatment D, Tiotropium 18 μg (Part 2)
- Sequence 2, Part 2 (Experimental): Period 1: Treatment B Period 2: Treatment C Period 3: Treatment A Period 4: Treatment D Period 5: Treatment E
  Interventions: Drug: Treatment A, AZD8871 dose A (Part 2); Drug: Treatment B, AZD8871 dose B (Part 2); Drug: Treatment C, Indacaterol 150 μg (Part 2); Drug: Treatment D, Tiotropium 18 μg (Part 2)
- Sequence 3, Part 2 (Experimental): Period 1: Treatment C Period 2: Treatment D Period 3: Treatment B Period 4: Treatment E Period 5: Treatment A
  Interventions: Drug: Treatment A, AZD8871 dose A (Part 2); Drug: Treatment B, AZD8871 dose B (Part 2); Drug: Treatment C, Indacaterol 150 μg (Part 2); Drug: Treatment D, Tiotropium 18 μg (Part 2)
- Sequence 4, Part 2 (Experimental): Period 1: Treatment D Period 2: Treatment E Period 3: Treatment C Period 4: Treatment A Period 5: Treatment B
  Interventions: Drug: Treatment A, AZD8871 dose A (Part 2); Drug: Treatment B, AZD8871 dose B (Part 2); Drug: Treatment C, Indacaterol 150 μg (Part 2); Drug: Treatment D, Tiotropium 18 μg (Part 2)
- Sequence 5, Part 2 (Experimental): Period 1: Treatment E Period 2: Treatment A Period 3: Treatment D Period 4: Treatment B Period 5: Treatment C
  Interventions: Drug: Treatment A, AZD8871 dose A (Part 2); Drug: Treatment B, AZD8871 dose B (Part 2); Drug: Treatment C, Indacaterol 150 μg (Part 2); Drug: Treatment D, Tiotropium 18 μg (Part 2)
- Sequence 6, Part 2 (Experimental): Period 1: Treatment D Period 2: Treatment C Period 3: Treatment E Period 4: Treatment B Period 5: Treatment A
  Interventions: Drug: Treatment A, AZD8871 dose A (Part 2); Drug: Treatment B, AZD8871 dose B (Part 2); Drug: Treatment C, Indacaterol 150 μg (Part 2); Drug: Treatment D, Tiotropium 18 μg (Part 2)
- Sequence 7, Part 2 (Experimental): Period 1: Treatment E Period 2: Treatment D Period 3: Treatment A Period 4: Treatment C Period 5: Treatment B
  Interventions: Drug: Treatment A, AZD8871 dose A (Part 2); Drug: Treatment B, AZD8871 dose B (Part 2); Drug: Treatment C, Indacaterol 150 μg (Part 2); Drug: Treatment D, Tiotropium 18 μg (Part 2)
- Sequence 8, Part 2 (Experimental): Period 1: Treatment A Period 2: Treatment E Period 3: Treatment B Period 4: Treatment D Period 5: Treatment C
  Interventions: Drug: Treatment A, AZD8871 dose A (Part 2); Drug: Treatment B, AZD8871 dose B (Part 2); Drug: Treatment C, Indacaterol 150 μg (Part 2); Drug: Treatment D, Tiotropium 18 μg (Part 2)
- Sequence 9, Part 2 (Experimental): Period 1: Treatment B Period 2: Treatment A Period 3: Treatment C Period 4: Treatment E Period 5: Treatment D
  Interventions: Drug: Treatment A, AZD8871 dose A (Part 2); Drug: Treatment B, AZD8871 dose B (Part 2); Drug: Treatment C, Indacaterol 150 μg (Part 2); Drug: Treatment D, Tiotropium 18 μg (Part 2)
- Sequence 10, Part 2 (Experimental): Period 1: Treatment C Period 2: Treatment B Period 3: Treatment D Period 4: Treatment A Period 5: Treatment E
  Interventions: Drug: Treatment A, AZD8871 dose A (Part 2); Drug: Treatment B, AZD8871 dose B (Part 2); Drug: Treatment C, Indacaterol 150 μg (Part 2); Drug: Treatment D, Tiotropium 18 μg (Part 2)

INTERVENTIONS:
Drug: Dose 1, AZD8871 50 μg (Part 1) — 50 µg of AZD8871 on Day 1; each dose of AZD8871 inhalation powder will be administered via single-dose dry powder inhaler (Genuair®)
  Arms: Sequence 1, Part 1; Sequence 3, Part 1; Sequence 4, Part 1
Drug: Dose 2, AZD8871 100 μg (Part 1) — 100 µg of AZD8871 on Day 1; each dose of AZD8871 inhalation powder will be administered via single-dose dry powder inhaler (Genuair®)
  Arms: Sequence 5, Part 1; Sequence 7, Part 1; Sequence 8, Part 1
Drug: Dose 3, AZD8871 300 μg (Part 1) — 300 µg of AZD8871 on Day 1; each dose of AZD8871 inhalation powder will be administered via single-dose dry powder inhaler (Genuair®)
  Arms: Sequence 1, Part 1; Sequence 2, Part 1; Sequence 4, Part 1
Drug: Dose 4, AZD8871 600 µg (Part 1) — 600 µg of AZD8871 on Day 1; each dose of AZD8871 inhalation powder will be administered via single-dose dry powder inhaler (Genuair®)
  Arms: Sequence 5, Part 1; Sequence 6, Part 1; Sequence 8, Part 1
Drug: Dose 5, AZD8871 1200 µg (Part 1) — 1200 µg of AZD8871 on Day 1; each dose of AZD8871 inhalation powder will be administered via single-dose dry powder inhaler (Genuair®)
  Arms: Sequence 1, Part 1; Sequence 2, Part 1; Sequence 3, Part 1
Drug: Dose 6, AZD8871 1800 μg (Part 1) — 1800 µg of AZD8871 on Day 1; each dose of AZD8871 inhalation powder will be administered via single-dose dry powder inhaler (Genuair®)
  Arms: Sequence 5, Part 1; Sequence 6, Part 1; Sequence 7, Part 1
Drug: Placebo, AZD8871 placebo (Part 1) — AZD8871 placebo on Day 1; each dose of AZD8871 placebo inhalation powder will be administered via single-dose dry powder inhaler (Genuair®)
  Arms: Sequence 2, Part 1; Sequence 3, Part 1; Sequence 4, Part 1; Sequence 6, Part 1; Sequence 7, Part 1; Sequence 8, Part 1
Drug: Treatment A, AZD8871 dose A (Part 2) — AZD8871 dose A once on Day 1; each dose of AZD8871 placebo inhalation powder will be administered via single-dose dry powder inhaler (Genuair®)
  Arms: Sequence 1, Part 2; Sequence 10, Part 2; Sequence 2, Part 2; Sequence 3, Part 2; Sequence 4, Part 2; Sequence 5, Part 2; Sequence 6, Part 2; Sequence 7, Part 2; Sequence 8, Part 2; Sequence 9, Part 2
Drug: Treatment B, AZD8871 dose B (Part 2) — AZD8871 dose B once on Day 1; each dose of AZD8871 placebo inhalation powder will be administered via single-dose dry powder inhaler(Genuair®)
  Arms: Sequence 1, Part 2; Sequence 10, Part 2; Sequence 2, Part 2; Sequence 3, Part 2; Sequence 4, Part 2; Sequence 5, Part 2; Sequence 6, Part 2; Sequence 7, Part 2; Sequence 8, Part 2; Sequence 9, Part 2
Drug: Treatment C, Indacaterol 150 μg (Part 2) — 150 μg of Indacaterol once on Day 1; each dose of Indacaterol dry inhalation powder will be administered via a dry powder inhaler (Onbrez Breezhaler®) as 1 hard capsule
  Arms: Sequence 1, Part 2; Sequence 10, Part 2; Sequence 2, Part 2; Sequence 3, Part 2; Sequence 4, Part 2; Sequence 5, Part 2; Sequence 6, Part 2; Sequence 7, Part 2; Sequence 8, Part 2; Sequence 9, Part 2
Drug: Treatment D, Tiotropium 18 μg (Part 2) — 18 μg of Tiotropium once on Day 1; each dose of Indacaterol dry inhalation powder will be administered via a dry powder inhaler (HandiHaler®) as 1 hard capsule
  Arms: Sequence 1, Part 2; Sequence 10, Part 2; Sequence 2, Part 2; Sequence 3, Part 2; Sequence 4, Part 2; Sequence 5, Part 2; Sequence 6, Part 2; Sequence 7, Part 2; Sequence 8, Part 2; Sequence 9, Part 2

SUMMARY:
This is a phase I, randomised, placebo-controlled 2-part study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD8871 delivered by inhalation, in asthmatic and chronic obstructive pulmonary disease (COPD) subjects.

DETAILED DESCRIPTION:
This study is an integrated Phase I protocol divided into 2 parts.

Part 1: single ascending dose study (6 AZD8871 dose levels) in 16 male subjects with mild asthma. AZD8871 will be administered (by the Genuair® inhaler) under supervision at the study centre, according to the randomisation scheme

Part 2: a 5 treatment period single dose study (of AZD8871 [two doses], indacaterol, tiotropium and placebo) in 40 male and non-childbearing female subjects with moderate to severe COPD. Each treatment period will be separated by a washout period of at least 7 days. The primary comparison for bronchodilation will be between AZD8871 doses and placebo.

ELIGIBILITY:
Inclusion Criteria:Part 1

1. Subjects who are able and willing to provide written informed consent prior to conducting any study-related procedures, including withdrawal of medications
2. Adult male subjects aged 18 to 70 years (both inclusive)
3. Body mass index (BMI) from 18 to 32 kg/m2 at screening
4. Clinical diagnosis of asthma (according to the Global Initiative for Asthma [GINA] guidelines) for at least 6 months prior to screening
5. Ability to change current asthma therapy, to discontinue previous prescribed medications after signature of informed consent as per required washout periods
6. Screening FEV1 value of ≥70% of the predicted normal value
7. FEV1 reversibility of ≥12% and an absolute increase of at least 200 mL over the baseline value within 30 min after inhalation of 400 µg (4 puffs) of salbutamol via a metered dose inhaler, with spacer device
8. Subjects using intermittent salbutamol and / or subjects on a stable dose of low dose Inhaled corticosteroid (as defined by the GINA guidelines) at least 4 weeks prior to screening
9. Predose FEV1 value of first treatment period within the range of ± 20% of the FEV1 measured at screening prior to salbutamol inhalation
10. No current smokers, no subjects with a smoking history during the last 12 months and no subjects with a total smoking history of more than 10 pack-years
11. No other relevant pulmonary disease or history of thoracic surgery
12. Subjects who are otherwise healthy as determined by medical history, physical examination, 12-lead ECG findings
13. Normal blood pressure (defined as Systolic blood pressure [SBP] between 100 and 140 mmHg for subjects ≤59 years of age and between 100 and 150 mmHg for subjects ≥60 years of age, and Diastolic blood pressure [DBP] between 40 and 90 mmHg) at screening
14. Subjects whose clinical laboratory test results are not clinically relevant and are acceptable to the Investigator.
15. Subjects who are negative for hepatitis B surface antigen (HBsAg), hepatitis B core (HBc) antibody (IgM), hepatitis C antibody and human immunodeficiency virus (HIV) I and II antibodies at screening
16. Subjects who are negative for drugs of abuse and alcohol tests at screening and admission
17. Subjects able to perform repeatable pulmonary function testing for FEV1 according to the American Thoracic Society (ATS) / European Respiratory Society (ERS) 2005(9) criteria at screening

Inclusion Criteria: Part 2

1. Adult male and non-childbearing female subjects aged ≥40 years with a clinical diagnosis of stable moderate to severe COPD according to GOLD guidelines at screening
2. Females must be of non-childbearing potential, confirmed at screening by fulfilling study predefined criteria
3. Post-salbutamol FEV1 <80% and ≥30% of the predicted normal value and post-salbutamol FEV1 / forced vital capacity (FVC) <70%
4. BMI < 40 kg/m2 at screening
5. Ability to change current COPD therapy, to discontinue previous prescribed medications after signature of informed consent as per required washout periods
6. Current or ex-smokers with a smoking history of ≥10 pack years
7. No evidence of clinically significant respiratory and / or cardiovascular conditions (e.g. uncontrolled hypertension) or laboratory abnormalities
8. No other relevant pulmonary disease or history of thoracic surgery
9. Subjects who are negative for HBsAg, HBc IgM, hepatitis C antibody and HIV I and II antibodies at screening
10. Subjects who are able and willing to provide written informed consent prior to conducting any study-related procedures, including withdrawal of medications
11. Medical history must be verified by either a personal physician or medical practitioner as appropriate
12. Subjects able to perform repeatable pulmonary function testing for FEV1 according to the ATS / ERS 2005(9) criteria at screening

Exclusion Criteria (Part 1 & 2):

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous enrolment or randomisation of treatment in the present study
3. Current evidence or recent history of any clinically significant and unstable disease (other than asthma/COPD) or abnormality that could put the subject at risk or could confound the results of the study
4. Subjects with a surgical history clinically relevant for the purpose of the study
5. History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localised basal cell carcinoma of the skin
6. Subjects with serious adverse reaction or serious hypersensitivity to Tiotropium (for Part 2 only), Indacaterol (for Part 2 only), or the formulation excipients (eg, lactose) or other drugs in the same pharmacologic class (for Part 1 and Part 2)
7. Current diagnosis of COPD (for Part 1 only) or history of / or current diagnosis for asthma (for Part 2 only)
8. Recent history of asthma / COPD exacerbation requiring hospitalisation or need for increased maintenance treatments for asthma / COPD within 6 weeks prior to screening or prior to randomisation
9. Use of daily oxygen therapy >10 h per day (for Part 2 only)
10. Use of systemic steroids for respiratory reasons within 6 weeks prior to screening
11. Lower respiratory tract infection within 6 weeks prior to screening or prior to randomisation
12. Upper respiratory tract infection requiring antibiotics within 6 weeks prior to screening or prior to randomisation
13. Current history of tuberculosis, bronchiectasis or other non-specific pulmonary disease
14. Subject with significant cardiovascular disease that may be vulnerable to cardiovascular instability
15. QTcF (QT interval corrected, Fridericia formula QT[msec]/RR[s]) interval, >450 ms for males and >470 ms for females at screening or prior to randomisation, or history of long QT syndrome
16. PR (duration in milliseconds from the beginning of wave P to onset of ventricular depolarisation [Q or R]) interval >200 ms at screening or prior to randomisation (for Part 1 only) Note: 4- 6 hours of ECG rhythm monitoring with telemetry will be performed on Day-1 to identify patients that may have any clinical significant abnormality prior to randomisation. If this occurs, patients should not participate in the study
17. Subjects with serum potassium concentration < 3.5mmol/l at screening
18. Subjects with a history of excessive use or abuse of alcohol within the past 2 years
19. Subjects with a history of drug abuse within the past 2 years
20. Subjects who are positive for drugs of abuse and alcohol tests at screening and prior to randomisation. Subjects consuming more than 14 (female subjects) or 21 (male subjects) units of alcohol a week
21. Donation or loss >400 ml of blood and plasma within the previous 3 months prior to screening
22. Subjects with a significant infection or known inflammatory process at screening or prior to randomisation
23. Subjects with acute gastrointestinal symptoms at the time of screening or prior to randomisation (eg, nausea, vomiting, diarrhoea, heartburn)
24. Subjects with an acute infection such as influenza at the time of screening or prior to randomisation
25. Male subjects who do not agree to follow instructions to avoid pregnancies
26. Subjects who are not able to adhere to the restrictions on prior and concomitant medications
27. Subjects who intend to use any concomitant medication not permitted by this protocol or who have not undergone the required washout period for a particular prohibited medication
28. Subjects who have used any investigational drug within 3 months prior to screening or within the equivalent time of 6 half-lives of receiving the last administration, whichever is longer
29. Subjects who have received the last dose of investigational product more than 3 months ago but who are on an extended follow-up
30. Subjects who are unlikely to co-operate with the requirements of the study, or the study center or the subjects who are unwilling or unable to follow the instructions of the principal investigator

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MBChB, MSc,MFPM, Principal Investigator — PAREXEL Early Phase Clinical Unit, London, United Kingdom; Dave Singh, Prof., Principal Investigator — The Medicines Evaluation Unit (MEU), Manchester, United Kingdom
Locations (2):
- United Kingdom (2):
  - Research Site, Harrow
  - Research Site, Manchester

REFERENCES:
- [Derived] Jimenez E, Astbury C, Albayaty M, Wahlby-Hamren U, Seoane B, Villarroel C, Pujol H, Bermejo MJ, Aggarwal A, Psallidas I. Navafenterol (AZD8871) in patients with mild asthma: a randomised placebo-controlled phase I study evaluating the safety, tolerability, pharmacokinetics, and pharmacodynamics of single ascending doses of this novel inhaled long-acting dual-pharmacology bronchodilator. Respir Res. 2020 Sep 9;21(Suppl 1):211. doi: 10.1186/s12931-020-01470-5. PMID 32907576
- [Derived] Singh D, Balaguer V, Astbury C, Wahlby-Hamren U, Jimenez E, Seoane B, Villarroel C, Lei A, Aggarwal A, Psallidas I. Navafenterol (AZD8871) in patients with COPD: a randomized, double-blind, phase I study evaluating safety and pharmacodynamics of single doses of this novel, inhaled, long-acting, dual-pharmacology bronchodilator. Respir Res. 2020 Sep 9;21(Suppl 1):102. doi: 10.1186/s12931-020-01347-7. PMID 32907566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 centres in the UK (one for each part). In part 1 of the study, the first patient was screened in October 2015 and the last patient visit was in March 2016. In part 2 of the study, the first patient was screened in April 2016 and the last patient visit was in August 2016.
Pre-assignment Details: 2-part study: Part 1: single ascending doses of AZD8871 (planned 50, 100, 300, 600, 1200, 1800 μg; actual dose 50, 200, 400, 900, 1800, 2100 μg) or placebo over 3 treatment periods; 2 cohorts (male; mild persistent asthma).
  Part 2: 5-way complete cross-over, single-dose; M/F, moderate/severe COPD; 2 doses of AZD8871, placebo, or 2 active controls.
Groups:
- Overall Population - Part 1: All individuals in Part 1 (patients who received single doses of AZD8871 [50, 400, 1800 μg for Cohort 1; 200, 900, 2100 μg for Cohort 2], or placebo, in 3 treatment periods separated by washout periods of 14 days).
- Overall Population - Part 2: All individuals involved in Part 2 (patients who received single doses of AZD8871 [400 and 1800 μg], placebo, indacaterol 150 μg, or tiotropium 18 μg, in 5 treatment periods separated by washout periods of 7-21 days.
Period: Treatment Period 1
Arm/Group | Overall Population - Part 1 | Overall Population - Part 2
Started | 16 | 38
Completed | 16 | 38
Not Completed | 0 | 0
Period: Washout Between Treatment Period 1 and 2
Arm/Group | Overall Population - Part 1 | Overall Population - Part 2
Started | 16 | 38
Completed | 16 | 33
Not Completed | 0 | 5
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 3
Period: Period 2
Arm/Group | Overall Population - Part 1 | Overall Population - Part 2
Started | 16 | 33
Completed | 16 | 33
Not Completed | 0 | 0
Period: Washout Between Treatment Period 2 and 3
Arm/Group | Overall Population - Part 1 | Overall Population - Part 2
Started | 16 | 33
Completed | 15 | 31
Not Completed | 1 | 2
Not completed — Sponsor's decision | 1 | 0
Not completed — Adverse Event | 0 | 2
Period: Period 3
Arm/Group | Overall Population - Part 1 | Overall Population - Part 2
Started | 15 | 31
Completed | 15 | 31
Not Completed | 0 | 0
Period: Washout Between Treatment Period 3 and 4
Arm/Group | Overall Population - Part 1 | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 31
Completed | 0 (Part 1 comprised 3 treatment periods only) | 29
Not Completed | 0 | 2
Not completed — Stability/variability criteria not met | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 4
Arm/Group | Overall Population - Part 1 | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 29
Completed | 0 (Part 1 comprised 3 treatment periods only) | 29
Not Completed | 0 | 0
Period: Washout Between Treatment Period 4 and 5
Arm/Group | Overall Population - Part 1 | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 29
Completed | 0 (Part 1 comprised 3 treatment periods only) | 28
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 5
Arm/Group | Overall Population - Part 1 | Overall Population - Part 2
Started | 0 (Part 1 comprised 3 treatment periods only) | 28
Completed | 0 (Part 1 comprised 3 treatment periods only) | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects who received at least 1 dose of the investigational product in Parts 1 and 2, respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | Overall Population - Part 1 | Overall Population - Part 2 | Total
Number analyzed (Participants) | 16 | 38 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (11.8) | 65.6 (6.4) | NA (NA) — Combined baseline demographic data were not calculated for Parts 1 and 2 of the study, which included separate patient populations (NA)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 16 | 16
  Male | 16 | 22 | 38

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Mild Persistent Asthma (Part 1) and COPD (Part 2) With at Least 1 Treatment-emergent Adverse Event
Description: An adverse event is the development of an undesirable medical condition, or the deterioration of a pre-existing medical condition, following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition can be symptoms, signs, or the abnormal results of laboratory parameters (haematology, blood chemistry, urinalysis, physical examination, 12-lead ECGs and telemetry, and vital signs). AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 18.1.
Time Frame: From the time of informed consent up to 14 (±2) days after the last dose of investigational product. Unresolved AEs were followed up by the investigator for as long as medically indicated.
Population: Safety population: all randomized subjects who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- AZD8871 50 μg (Part 1); AZD8871 200 μg (Part 1); AZD8871 400 μg (Part 1); AZD8871 900 μg (Part 1); AZD8871 1800 μg (Part 1); AZD8871 2100 μg (Part 1); Placebo (Part 1); AZD8871 400 μg (Part 2); AZD8871 1800 μg (Part 2); Placebo (Part 2): Single-dose, oral inhalation by Genuair® single-dose dry powder inhaler (DPI)
- Indacaterol 150 μg (Part 2): Single-dose, oral inhalation by Onbrez Breezhaler® single-dose dry powder inhaler (DPI)
- Tiotropium 18 μg (Part 2): Single-dose, oral inhalation by HandiHaler® single-dose dry powder inhaler (DPI)
Arm/Group | AZD8871 50 μg (Part 1) | AZD8871 200 μg (Part 1) | AZD8871 400 μg (Part 1) | AZD8871 900 μg (Part 1) | AZD8871 1800 μg (Part 1) | AZD8871 2100 μg (Part 1) | Placebo (Part 1) | AZD8871 400 μg (Part 2) | AZD8871 1800 μg (Part 2) | Indacaterol 150 μg (Part 2) | Tiotropium 18 μg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 12 | 34 | 31 | 32 | 30 | 32
Participants | 5 | 5 | 3 | 3 | 3 | 2 | 7 | 18 | 7 | 12 | 11 | 11

2. Primary Outcome: Number of Participants With Clinically Relevant Abnormalities in Blood Pressure
Description: Blood pressure (BP) measurements (diastolic [DBP] and systolic BP [SBP]) taken after ~5 minutes rest in supine position, at screening, baseline (≤1 hour before IP administration), 10 and 30 minutes, 1, 2, 3, 4, 8, 12 hours (Day 1) and 24 and 36 hours (Day 2) after IP administration. Normal BP at screening: SBP 100-140 mmHg (subjects aged ≤59 years) and 100-150 mmHg (subjects aged ≥60 years), and DBP 40-90 mmHg.
  Criteria for notable changes in BP:
  High SBP: (≥180 and increase over baseline (predose) ≥20) or (≥200 and baseline <200) Low SBP: (≤ 90 and decrease over baseline ≥20) or (≤75 and baseline >75) High DBP: (≥105 and increase over baseline ≥15) or (≥115 and baseline <115) Low DBP: (≤50 and decrease over baseline ≥15) or (≤40 and baseline >40) All out of range values were flagged to the principal investigator who assessed clinical relevance based on medical criteria at individual subject level. Clinically relevant findings were assessed until considered non-clinically relevant.
Time Frame: From the time of informed consent up to 36 hours after last dose of IP.
Population: Safety population: all randomized subjects who received at least 1 dose of the investigational product
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8871 50 μg (Part 1) | AZD8871 200 μg (Part 1) | AZD8871 400 μg (Part 1) | AZD8871 900 μg (Part 1) | AZD8871 1800 μg (Part 1) | AZD8871 2100 μg (Part 1) | Placebo (Part 1) | AZD8871 400 μg (Part 2) | AZD8871 1800 μg (Part 2) | Indacaterol 150 μg (Part 2) | Tiotropium 18 μg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 12 | 34 | 31 | 32 | 30 | 32
Participants | 0 (8.7) | 0 (2.1) | 0 (4.3) | 0 (7.2) | 0 (3.4) | 0 (11.7) | 0 (5.7) | 0 (8.3) | 0 (4.5) | 0 (6.3) | 0 (6.8) | 0 (9.6)

3. Primary Outcome: Number of Participants With Clinically Relevant Abnormalities in Electrocardiograms (HR, QTcF and Other ECG Parameters).
Description: HR, QTcF and other ECG abnormalities were assessed by local digital 12-lead ECG performed in triplicate at the time points indicated:
  ECG (Parts 1 and 2) was assessed at Screening, Day 1 baseline, 10 min, 30 min, 1 hour (h), 2 h, 3 h, 4 h, 8 h, 12 h, 24 h, 36 h after dosing.
  Telemetry (Part 1), assessed with at least 2 lead real time display, was recorded at Day -1 (4-6 hours continuous recording, at the time this was more convenient for the logistics of the unit) and on Day 1 from the time of the IP administration up to at least 24 hours, but if advised by the Investigator or designee, then up to 36 hours after IP administration.
  Abnormal findings were flagged to the principal investigator who assessed clinical relevance based on medical criteria at individual subject level. Clinically relevant findings were assessed until the abnormality was considered non-clinically relevant.
Time Frame: From the time of informed consent up to 36 hours after last dose of IP.
Population: Safety population: all randomized subjects who received at least 1 dose of the investigational product
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8871 50 μg (Part 1) | AZD8871 200 μg (Part 1) | AZD8871 400 μg (Part 1) | AZD8871 900 μg (Part 1) | AZD8871 1800 μg (Part 1) | AZD8871 2100 μg (Part 1) | Placebo (Part 1) | AZD8871 400 μg (Part 2) | AZD8871 1800 μg (Part 2) | Indacaterol 150 μg (Part 2) | Tiotropium 18 μg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 12 | 34 | 31 | 32 | 30 | 32
Participants | 0 (4.5) | 0 (3.9) | 0 (3.7) | 0 (3.2) | 0 (5.2) | 0 (4.8) | 0 (6.2) | 0 (6.2) | 0 (7.7) | 0 (5.5) | 0 (4.7) | 0 (6.1)

4. Primary Outcome: Number of Participants With Clinically Relevant Abnormalities in Clinical Biochemistry, Hematology and Urinalysis
Description: A composite of clinically relevant abnormalities in clinical biochemistry, hematology and urinalysis laboratory evaluations. Laboratory tests (haematology, blood chemistry, and urinalysis) were performed at screening, at Day -1 (Part 1 only), at 24 hours (Day 2) and at follow-up (7 [±2] days) after IP administration. Coagulation was only performed at screening; TSH, T4 only at screening, at Day-1 and at follow-up.
  Abnormal findings were flagged to the principal investigator who assessed clinical relevance based on medical criteria at individual subject level. Clinically relevant findings were assessed until the abnormality was considered non-clinically relevant.
Time Frame: From the time of informed consent up to 7 days after the last dose of IP.
Population: Safety population: all randomized subjects who received at least 1 dose of the investigational product
Measure: Count of Participants; unit: Participants
Arm/Group | AZD8871 50 μg (Part 1) | AZD8871 200 μg (Part 1) | AZD8871 400 μg (Part 1) | AZD8871 900 μg (Part 1) | AZD8871 1800 μg (Part 1) | AZD8871 2100 μg (Part 1) | Placebo (Part 1) | AZD8871 400 μg (Part 2) | AZD8871 1800 μg (Part 2) | Indacaterol 150 μg (Part 2) | Tiotropium 18 μg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 12 | 34 | 31 | 32 | 30 | 32
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) on Day 2
Description: Pharmacodynamics of AZD8871 before (-45 min and -15 min pre-dose) and after single dosing of AZD8871 Forced expiratory volume in 1 second (FEV1) on Day 2 (defined as the average of the values 23:00 and 24:00 hours after the morning dose of investigational product)
Time Frame: Baseline (Day 1) to 36 hours post-dose (Day 2)
Population: The PP population is defined as all randomised subjects who satisfied the main I/E criteria, received IP, completed at least 1 treatment period, and did not present major violations to the protocol
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | AZD8871 50 μg (Part 1) | AZD8871 200 μg (Part 1) | AZD8871 400 μg (Part 1) | AZD8871 900 μg (Part 1) | AZD8871 1800 μg (Part 1) | AZD8871 2100 μg (Part 1) | Placebo (Part 1) | AZD8871 400 μg (Part 2) | AZD8871 1800 μg (Part 2) | Indacaterol 150 μg (Part 2) | Tiotropium 18 μg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 12 | 34 | 31 | 32 | 30 | 32
Liters | -0.0375 (0.3449) | 0.2183 (0.1631) | 0.2883 (0.1418) | 0.1858 (0.3528) | 0.3275 (0.0708) | 0.4630 (0.2065) | -0.0600 (0.3099) | 0.0738 (0.1212) | 0.1731 (0.1761) | 0.1036 (0.1286) | 0.1055 (0.1922) | -0.0294 (0.0768)
Statistical Analysis 1: Comparison: AZD8871 400 μg (Part 2) vs Placebo (Part 2); Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Square Mean = 0.111, 95% CI 2-sided [0.0585 to 0.163], Standard Error of Mean 0.0265
Statistical Analysis 2: Comparison: AZD8871 1800 μg (Part 2) vs Placebo (Part 2); Test type: Superiority or Other; p < 0.0001, ANCOVA; Least square mean = 0.210, 95% CI [0.156 to 0.264], Standard Error of Mean 0.0272

6. Secondary Outcome: Cmax of AZD8871 in Parts 1 and 2
Description: Cmax (maximum observed plasma drug concentrations) of AZD8871 on Day 1 of each treatment period.
Time Frame: Pre-dose, and 5 min, 15 min, 30 min, 45 min, 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h (Day 1), 24 h, and 36 h (Day 2) post-dose
Population: Pharmacokinetic population: defined as all randomised subjects who have received at least 1 dose of investigational product in at least 1 treatment period and have evaluable PK parameters. AZD8871 plasma PK assessed following dosing with AZD8871 only (not placebo, indacaterol, or tiotropium).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | AZD8871 50 μg (Part 1) | AZD8871 200 μg (Part 1) | AZD8871 400 μg (Part 1) | AZD8871 900 μg (Part 1) | AZD8871 1800 μg (Part 1) | AZD8871 2100 μg (Part 1) | Placebo (Part 1) | AZD8871 400 μg (Part 2) | AZD8871 1800 μg (Part 2) | Indacaterol 150 μg (Part 2) | Tiotropium 18 μg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 0 | 18 | 15 | 0 | 0 | 0
pg/mL | 34.77 (60.77) | 174.1 (43.74) | 313.4 (46.56) | 797.3 (20.99) | 1351 (20.32) | 1243 (24.33) |  | 199.3 (37.40) | 810.8 (36.59) |  |  |

7. Secondary Outcome: Tmax of AZD8871 in Parts 1 and 2
Description: tmax (time to reach maximum concentration) of AZD8871 on Day 1 of each treatment period.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: Hours
Arm/Group | AZD8871 50 μg (Part 1) | AZD8871 200 μg (Part 1) | AZD8871 400 μg (Part 1) | AZD8871 900 μg (Part 1) | AZD8871 1800 μg (Part 1) | AZD8871 2100 μg (Part 1) | Placebo (Part 1) | AZD8871 400 μg (Part 2) | AZD8871 1800 μg (Part 2) | Indacaterol 150 μg (Part 2) | Tiotropium 18 μg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 0 | 18 | 15 | 0 | 0 | 0
Hours | 0.88 [0.52 to 1.03] | 0.86 [0.48 to 1.00] | 1.00 [0.75 to 1.05] | 1.00 [0.98 to 1.02] | 1.49 [0.73 to 2.03] | 1.02 [1.00 to 2.00] |  | 1.00 [0.75 to 3.00] | 2.00 [0.75 to 3.00] |  |  |

8. Secondary Outcome: AUC(0-t) of AZD8871 in Parts 1 and 2
Description: AUC(0-t) (area under the concentration-time curve from time zero to time of the last quantifiable measurable concentration) of AZD8871 on Day 1 of each treatment period.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | AZD8871 50 μg (Part 1) | AZD8871 200 μg (Part 1) | AZD8871 400 μg (Part 1) | AZD8871 900 μg (Part 1) | AZD8871 1800 μg (Part 1) | AZD8871 2100 μg (Part 1) | Placebo (Part 1) | AZD8871 400 μg (Part 2) | AZD8871 1800 μg (Part 2) | Indacaterol 150 μg (Part 2) | Tiotropium 18 μg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 0 | 16 | 15 | 0 | 0 | 0
pg*h/mL | 110 (69.17) | 631.3 (30.40) | 1397 (31.41) | 3299 (27.00) | 6055 (24.98) | 6418 (35.13) |  | 1239 (37.70) | 6159 (44.30) |  |  |

9. Secondary Outcome: AUC(0-24) of AZD8871 in Parts 1 and 2
Description: AUC(0-24) (area under the concentration-time curve from zero to 24h) of AZD8871 on Day 1 of each treatment period.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | AZD8871 50 μg (Part 1) | AZD8871 200 μg (Part 1) | AZD8871 400 μg (Part 1) | AZD8871 900 μg (Part 1) | AZD8871 1800 μg (Part 1) | AZD8871 2100 μg (Part 1) | Placebo (Part 1) | AZD8871 400 μg (Part 2) | AZD8871 1800 μg (Part 2) | Indacaterol 150 μg (Part 2) | Tiotropium 18 μg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 0 | 18 | 15 | 0 | 0 | 0
pg*h/mL | 118.9 (60.19) | 567.9 (29.74) | 1265 (32.44) | 3020 (25.71) | 5587 (25.40) | 5922 (34.32) |  | 1195 (38.91) | 5659 (43.68) |  |  |

10. Other Pre Specified Outcome: AUC of AZD8871 in Parts 1 and 2
Description: AUC (area under the concentration-time curve from time 0 to infinity) of AZD8871 on Day 1 of each treatment period
Time Frame: Predose, and 5 min, 15 min, 30 min, and 45 min, at 1 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h (Day 1), 24 h and 36 h (Day 2) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | AZD8871 50 μg (Part 1) | AZD8871 200 μg (Part 1) | AZD8871 400 μg (Part 1) | AZD8871 900 μg (Part 1) | AZD8871 1800 μg (Part 1) | AZD8871 2100 μg (Part 1) | Placebo (Part 1) | AZD8871 400 μg (Part 2) | AZD8871 1800 μg (Part 2) | Indacaterol 150 μg (Part 2) | Tiotropium 18 μg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5 | 0 | 18 | 15 | 0 | 0 | 0
pg*h/mL | 123.1 (75.48) | 774.5 (32.64) | 1671 (28.54) | 3831 (28.72) | 6941 (22.23) | 7164 (34.10) |  | 1459 (39.19) | 6769 (44.65) |  |  |

11. Other Pre Specified Outcome: Elimination Half-life of AZD8871 in Parts 1 and 2
Description: Elimination half-life (t½λz) for AZD8871 on Day 1 of each treatment period. t½λz was generally calculated over a period of less than 3 times the resultant half-life
Time Frame: as for outcome 10
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | AZD8871 50 μg (Part 1) | AZD8871 200 μg (Part 1) | AZD8871 400 μg (Part 1) | AZD8871 900 μg (Part 1) | AZD8871 1800 μg (Part 1) | AZD8871 2100 μg (Part 1) | Placebo (Part 1) | AZD8871 400 μg (Part 2) | AZD8871 1800 μg (Part 2) | Indacaterol 150 μg (Part 2) | Tiotropium 18 μg (Part 2) | Placebo (Part 2)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 0 | 18 | 15 | 0 | 0 | 0
Hours | 9.439 (7.350) | 23.10 (2.809) | 20.81 (5.384) | 18.86 (3.959) | 19.29 (5.468) | 15.96 (2.789) |  | 14.20 (5.521) | 12.89 (2.268) |  |  |

ADVERSE EVENTS:
Time Frame: From the time of informed consent up to 14 (±2) days after the last dose of investigational product (IP). Treatment-emergent adverse events were those reported after the first dose of IP up to 14 (±2) days after the last dose of IP. Unresolved AEs were followed up by the investigator for as long as medically indicated.
Description: The Safety population comprised all randomised subjects who received at least 1 dose of the IP.
Arm/Group | AZD8871 50 μg (Part 1) | AZD8871 200 μg (Part 1) | AZD8871 400 μg (Part 1) | AZD8871 900 μg (Part 1) | AZD8871 1800 μg (Part 1) | AZD8871 2100 μg (Part 1) | Placebo (Part 1) | AZD8871 400 μg (Part 2) | AZD8871 1800 μg (Part 2) | Indacaterol 150 μg (Part 2) | Tiotropium 18 μg (Part 2) | Placebo (Part 2)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/12 | 1/34 | 0/31 | 0/32 | 1/30 | 0/32
Other Adverse Events (participants affected / at risk) | 5/6 | 5/6 | 3/6 | 3/6 | 3/6 | 2/5 | 12/12 | 8/34 | 4/31 | 6/32 | 8/30 | 8/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8871 50 μg (Part 1) (N=6) | AZD8871 200 μg (Part 1) (N=6) | AZD8871 400 μg (Part 1) (N=6) | AZD8871 900 μg (Part 1) (N=6) | AZD8871 1800 μg (Part 1) (N=6) | AZD8871 2100 μg (Part 1) (N=5) | Placebo (Part 1) (N=12) | AZD8871 400 μg (Part 2) (N=34) | AZD8871 1800 μg (Part 2) (N=31) | Indacaterol 150 μg (Part 2) (N=32) | Tiotropium 18 μg (Part 2) (N=30) | Placebo (Part 2) (N=32)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Physical assault (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8871 50 μg (Part 1) (N=6) | AZD8871 200 μg (Part 1) (N=6) | AZD8871 400 μg (Part 1) (N=6) | AZD8871 900 μg (Part 1) (N=6) | AZD8871 1800 μg (Part 1) (N=6) | AZD8871 2100 μg (Part 1) (N=5) | Placebo (Part 1) (N=12) | AZD8871 400 μg (Part 2) (N=34) | AZD8871 1800 μg (Part 2) (N=31) | Indacaterol 150 μg (Part 2) (N=32) | Tiotropium 18 μg (Part 2) (N=30) | Placebo (Part 2) (N=32)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (6) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 5 (5) | 3 (4) | 4 (4) | 7 (7) | 7 (7)
Chronic obstructive pulmonary disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the Principal Investigator (PI) will be subject to mutual agreement between the PI and the sponsor.